CLINICAL TRIAL: NCT06304831
Title: Facility Ratings to Improve Satisfaction With Heath Care for Children
Brief Title: Use of Facility Ratings to Improve Satisfaction With Heath Care for Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Lao Tropical and Public Health Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SwissTI
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-03

CONDITIONS: Quality of Health Care

STUDY DESIGN:
Intervention Model Description: This study consists of a randomized controlled experiment involving 660 mothers with children less than 2 years old. Participants will be randomly assigned to one of two groups: 1) a control group that will not receive any information about providers and 2) an intervention group that will receive biweekly updates about quality ratings based on reviews collected from mothers of young children in the study areas. The unit of randomization will be the individual participant. A simple random number draw generated by the ODK package installed on the tablets will be used to assign participants to treatment and control with equal probability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive biweekly updates about quality ratings of recently visited health care providers for children by everyone enrolled in the study.
  Interventions: Behavioral: Quality ratings of health care providers for children
- Control (No Intervention): The control group will not receive any information about health care providers for children.

INTERVENTIONS:
Behavioral: Quality ratings of health care providers for children — Ratings of overall and components of quality (provider knowledge, respectfulness of provider, respectfulness of staff, cleanliness, cost) of health care providers for children will be provided on a webpage. The webpage will be updated every week and participants will be invited to access the latest ratings biweekly.
  Arms: Intervention

SUMMARY:
Despite increasing options for public and private health care providers in Laos, choosing a high-quality health provider or a facility is difficult because timely and reliable information about providers is not readily available. People rely on social networks or previous experiences to select providers. However, in Laos, only 28% describe their recent visit to a health care provider as high-quality suggesting that while there are increasing options for care, people may need support to find providers that meet their quality needs. Rapid adoption of mobile phones in Laos, particularly in urban areas, offer opportunities to enhance people's access to timely quality information about health care providers. The study team will use mobile phones to collect and disseminate quality information about providers - known to be valued by Laotians - to improve their access to quality care as well as their overall satisfaction with care.

DETAILED DESCRIPTION:
While access to health care is expanding globally, there is appreciable variation in the quality of care among providers with low-quality care accounting for up-to 5 million deaths each year. These numbers are expected to grow as more people seek care and as the burden of disease shifts to complex conditions.

Expanding access has also resulted in increasing options for public and private health care providers. Selecting a health provider or a facility, however, is difficult because timely and reliable information about providers is not readily available. People often rely on social networks or previous experiences to select providers. However, in Lao PDR, only 28% describe their recent visit to a health care provider as high-quality, suggesting that while there are increasing options for care, people may need support to find providers that meet their quality needs.

In order to inform efforts to improve people's access to high-quality care, there is a need for evidence on mechanisms to empower people to identify and use high-quality care. In LMICs, majority of efforts to date has focused on supply-side efforts. While there are new initiatives to study population perspectives and people's care experiences, measures to "ignite demand" for high-quality care are not well understood.

The investigators plan to conduct a randomized-controlled experiment using mobile-phones to study whether routinely collected information on quality of care received by peers can improve access to high-quality care and patient satisfaction. The investigators plan to study whether participants switched providers based on the information provided and the type of information mothers used to switch providers. Additionally, The investigators plan to study whether information about providers led women to be more satisfied with health care services for their child or children. Study participants will include mothers living in an urban setting with less than 2-year old children and already enrolled in an on-going VITERBI cohort in Vientiane, the capital city.

ELIGIBILITY:
Inclusion Criteria:

* All women 18 years of age and older and enrolled in Vientiane Multigenerational Birth Cohort (VITERBI) with at least one child less than two years old, able to read, have exclusive access to a mobile phone, have a WhatsApp account, understand and sign the ICF will be eligible to participate in the study. The eligibility criteria will be assessed using data collected from VITERBI. Ability to read will be tested using a script in Lao, "I use my mobile phone every day."

Exclusion Criteria:

* Eligible women unwilling to sign informed consent, without exclusive access to a mobile phone, unable to read the test script, or unable operate a mobile phone will be excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 559 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-10-23 (Actual)

PRIMARY OUTCOMES:
Proportion of mothers that change their preferred health care providers for children for non-urgent care | 3 months
  The primary outcome of this study is the proportion of mothers that changed their preferred health care facility for non-urgent child care services between baseline and endline surveys. Non-urgent care is defined as children with mild fever of 38 degrees along with cough. During the baseline and endline surveys, participants will be asked to specify their preferred location for non-urgent child care as follows: "If your child is sick tomorrow with mild fever of 38 degrees Celsius and cough, which hospital, clinic or health center will you take your child to?" The primary outcome will be a binary indicator for participants changing their preferred location between baseline and endline.

SECONDARY OUTCOMES:
Proportion of mothers satisfied with health care for their children of their most recent visit | 3 months
  The secondary outcome measure will be satisfaction with the health care facility visited most recently for care for their child under age 2. This measure will only be available for mothers seeking care for their child during the study period. This will be a binary variable and satisfaction will be defined as answering "Excellent" or "Very good" (instead of "Good", "Fair", or "Poor") to the question, "How would you rate the overall quality of care you received?", referring to the most recent visit for their child under age 2 within the past 3 months.
Number and type of health care providers used in the past 3 months | 3 months
  This secondary outcome is the number and types of providers (government health centers, government hospitals, private clinics and private hospitals) visited by mothers for health care for their children during the study period. Every 2 weeks, all enrolled participants will be asked: "Did you visit a health center, hospital or clinic for child in the last two weeks?" using a mobile application. Ones that respond "Yes," will be requested to complete an online survey about the visit, which will ask them to specify the health facility visited.
Proportion of mothers that change their most recently visited health care providers for children | 3 months
  This secondary outcome is the proportion of mothers that changed the most recently visited health care facility for child care services between baseline and endline surveys. This measure will be a binary variable and will only be available for caregivers using care both within the three months periods preceding the baseline and endline survey.
Proportion of mothers choosing the preferred facility for non-urgent care because of online or digital information sources | 3 months
  This secondary outcome is the proportion of mothers that used online or digital information sources reasons for choosing providers for non-urgent care. During the baseline and endline surveys, participants will be asked to specify their preferred location for non-urgent child care as follows: "If your child is sick tomorrow with mild fever of 38 degrees Celsius and cough, which hospital, clinic or health center will you take your child to?" After this question, participants will be asked, "Was this choice informed by online or digital information services?" This outcome will be a binary variable.
Proportion of mothers that change their preferred health care providers for children for urgent care | 3 months
  This secondary outcome is the proportion of mothers that changed their preferred health care facility for urgent child care services between baseline and endline surveys. Urgent care is defined as children with high fever and a red rash covering their body. During the baseline and endline surveys, participants will be asked to specify their preferred location for urgent child care as follows: "If your child is sick tomorrow with a very high fever of 39-40 degrees and a red rash covering their body, which hospital, clinic or health center will you take your child to?" This outcome will be a binary indicator for participants changing their preferred location for urgent care between baseline and endline.
Proportion of mothers confident they can identify the best place for getting care for sick children | 3 months
  This secondary outcome is the proportion of mothers can identify the best place for getting care for sick children based on his/her health problems. During the baseline and endline surveys, all participants will be asked to respond with "Strongly agree," "Agree," "Unsure," "Disagree" or "Strongly disagree" to the following question: "I am able to identify the best place to get care for my child when he/she is sick." This outcome will be a binary variable. Participants responding with "Strongly Agree" or "Agree" will be defined as being confident that they can identify the best place for getting care for sick children and participants responding with "Unsure," "Disagree," or "Strongly Disagree" will be defined as not being confident where to seek care.

CONTACTS AND LOCATIONS:
Overall Officials: Günther Fink, PhD, Study Chair — Swiss Tropical & Public Health Institute; Amit Aryal, MPH, Principal Investigator — Swiss Tropical & Public Health Institute
Locations (1):
- Lao Tropical and Public Health Institute, Vientiane, Vientiane Capital, Laos

IPD SHARING:
Plan to Share IPD: No
De-identified survey data will be retained for at least 15 years on a public data repository after publication of study findings.

REFERENCES:
- [Derived] Aryal A, Clarke-Deelder E, Sayasone S, Fink G. Informing Facility Selection Through a Web-Based User Ratings System: Protocol for a Randomized Controlled Trial Among Mothers in Urban Lao People's Democratic Republic. JMIR Res Protoc. 2025 Sep 4;14:e66085. doi: 10.2196/66085. PMID 40907019